CLINICAL TRIAL: NCT05789628
Title: A Look at the Patterns in Medical Research Participation Among Patients With Cervical Cancer
Brief Title: Discovering Factors in Cervical Cancer Patients' Clinical Trial Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 85789149
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The percentages of participants in clinical studies haven't always been perfectly representative of a particular group.

This research examines the variables that affect a patient's choice to enroll in, discontinue participation in, or resume participation in a clinical trial for cervical cancer.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future cervical cancer studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Ability to understand and the willingness to sign a written informed consent document.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who are actively considering involvement in an observational cervical cancer clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a cervical cancer clinical study. | 3 months
Number of cervical cancer study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hu L, Bell D, Antani S, Xue Z, Yu K, Horning MP, Gachuhi N, Wilson B, Jaiswal MS, Befano B, Long LR, Herrero R, Einstein MH, Burk RD, Demarco M, Gage JC, Rodriguez AC, Wentzensen N, Schiffman M. An Observational Study of Deep Learning and Automated Evaluation of Cervical Images for Cancer Screening. J Natl Cancer Inst. 2019 Sep 1;111(9):923-932. doi: 10.1093/jnci/djy225. PMID 30629194
- [Background] Peirson L, Fitzpatrick-Lewis D, Ciliska D, Warren R. Screening for cervical cancer: a systematic review and meta-analysis. Syst Rev. 2013 May 24;2:35. doi: 10.1186/2046-4053-2-35. PMID 23706117
- [Background] Saei Ghare Naz M, Kariman N, Ebadi A, Ozgoli G, Ghasemi V, Rashidi Fakari F. Educational Interventions for Cervical Cancer Screening Behavior of Women: A Systematic Review. Asian Pac J Cancer Prev. 2018 Apr 25;19(4):875-884. doi: 10.22034/APJCP.2018.19.4.875. PMID 29693331

DOCUMENTS (1):
  • Informed Consent Form (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT05789628/ICF_000.pdf